CLINICAL TRIAL: NCT07099976
Title: PromotIng Optimal Treatment for Community-acquired PNeumonia in EmErgency Rooms (PIONEERS): a Multicentre, Randomized, Open-labelled, Controlled, Clinical Trial
Brief Title: PromotIng Optimal Treatment for Community-acquired PNeumonia in EmErgency Rooms
Acronym: PIONEERS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jeffrey (Other)
Responsible Party: Sponsor-Investigator, Jeffrey, Associate Professor, McMaster University
Organization: McMaster University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 5063-CTIA-Mar/2025-118722
Record Dates: First submitted 2025-04-28; First posted 2025-08-01 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Community-Acquired Pneumonia (CAP); Pneumonia
Keywords: Pneumonia; Antibiotics
MeSH Terms: conditions — Community-Acquired Pneumonia; Pneumonia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The novel care pathway intervention (Experimental): The novel care pathway intervention will incorporate multiple factors to determine risk of bacterial CAP. At recruitment, POC CRP testing, and bioMérieux Spotfire testing of nasopharyngeal swabs (NPS) will identify those who are at appreciable risk and will receive a prescription for antibiotic treatment on day 0. Please refer to the Specimen Collection and Processing manual for more specific information on the collection process. Appreciable-risk participants will be referred back to the clinical team to be given amoxicillin, the current standard of care in Canada (those with penicillin allergy will presumably receive an appropriate substitution as per local guidelines). Low-risk participants will be discharged home without antibiotics.
  Interventions: Diagnostic Test: The novel care pathway intervention
- Control Group (Active Comparator): Participants will be recruited in the ED and will be managed as per the treating clinician; the study team will not influence management
  Interventions: Other: Usual Care Alone

INTERVENTIONS:
Diagnostic Test: The novel care pathway intervention — The pathway uses already-ascertained data, bioMérieux Spotfire testing, and POC CRP testing to stratify patients into risk categories. The first step in the pathway will be POC CRP testing; children with CRP > 60 mg/L will be deemed 'appreciable risk', whereas those with CRP < 20 mg/L will be deemed 'low risk'. The CRP cut-offs of 20mg/L (more sensitive) and 60mg/L (more specific) were selected after reviewing the literature, with particular emphasis on meta-analyses; other large recent studies have also used 60mg/L as an upper cut-off for bacterial infection. Participants with CRP between 20-60mg/L will be categorized further to identify children either more likely to have bacterial pneumonia or more intolerant of misclassification. 'If they have O2 saturation <95% AND tachypnoea as per age-specific norms, they will be 'appreciable risk' (>60 bpm for age <1 y, >50 bpm for 1-2 y, >40 bpm for 2-4 y, and >30 bpm for >4 y).
  Arms: The novel care pathway intervention
Other: Usual Care Alone — Participants will be recruited in the ED and will be managed as per the treating clinician; the study team will not influence management.
  Arms: Control Group

SUMMARY:
In North America, up to 5% of preschoolers develop community-acquired pneumonia (CAP) every year. Pneumonia is the second-leading reason for paediatric hospitalization in both Canada and the US; approximately 20% of children hospitalized with CAP may need intensive care, which can result in significant morbidity. Given this burden of disease, it is critical that CAP is managed appropriately. Specific therapy for CAP is dependent on microbiologic aetiology, as bacterial disease will improve with antibiotic treatment.

DETAILED DESCRIPTION:
Unfortunately, there are no features on history or physical examination that are highly specific for either viral or bacterial disease. Although bacterial disease is more often associated with consolidations, validated radiographic criteria for reliably distinguishing between viral and bacterial pneumonia do not exist. Furthermore, children, unlike adults, commonly develop viral pneumonia or bacterial-viral coinfections; one large prospective study of children hospitalized with CAP in the USA reported that 66% had a respiratory virus detected and 26% had proven coinfections. Consequently, though physicians are aware that antibiotics do not improve the course of children with viral illnesses, the inability to reliably discriminate between viral and bacterial disease results in the vast majority of children with even non-severe CAP (ie. that can be managed as an outpatient) receiving antibiotics. This may be because clinicians are not aware how much paediatric CAP is viral, but is probably also related to physician beliefs/attitudes. These include the desire to be 'safe', the belief that families want antibiotics, and the perception that it is easier and quicker to prescribe than to explain why antibiotics are not required.

Minimizing inappropriate antimicrobial prescribing is an important strategy to prevent further emergence of circulating antimicrobial resistance. The WHO's Global Action Plan on Antimicrobial Resistance states that 'evidence-based prescribing should be the standard of care'. Optimizing antimicrobial prescribing, also known as 'antimicrobial stewardship', is the main strategy to deal with escalating antimicrobial resistance and has been called 'a fiduciary responsibility for all healthcare institutions across the continuum of care'. Antibiotic stewardship is critical to reducing the dramatic increase in antimicrobial resistance seen in Canada and worldwide, which is why CIHR continues to encourage antimicrobial stewardship research. The Public Health Agency of Canada's 2023 Pan-Canadian Action Plan on Antimicrobial Resistance explicitly calls for research to 'support the development and uptake of diagnostics…that support antimicrobial stewardship, including point-of-care tools'. Antimicrobials routinely prescribed to children can produce problematic side effects and impact normal microbiota, which can influence the development of obesity, atopy, and other disorders.

It has now been definitively established that short course (3-5 day) antibiotic treatment is equally effective as longer courses of antibiotics for non-severe paediatric CAP. The investigators conducted the first of these trials to be published, a multi-year RCT at McMaster Children's Hospital (MCH) and the Children's Hospital of Eastern Ontario (CHEO), enrolling children with non-severe CAP, randomizing to either 5 or 10 days of amoxicillin (duration blinded using placebos), and demonstrated that clinical response at 14-21 days was comparable between groups. Shortening durations further would not seem advisable, given that one trial in Israel found more failures in children given 3 days of antibiotics and that it has been shown that 3 days of antibiotics is superior to placebo for the treatment of paediatric CAP. The investigators believe a better strategy would be to determine how to better identify children with purely viral disease, given that these cases represent the majority of paediatric CAP, and/or enable front-line clinicians to more effectively withhold antibiotics entirely from children at lower risk of bacterial disease. (The investigators note that in these referenced randomized trials and systematic reviews, antibiotic treatment was not associated with large improvements in cure rates; this probably speaks to the fact that only a small proportion of paediatric CAP is bacterial, as reliable discrimination between viral and bacterial disease is not possible on clinical grounds.)

There have been efforts to use biomarkers alone to improve prescribing for respiratory infections. One systematic review found that point-of-care C-reactive protein (POC CRP) testing was associated with significantly decreased antibiotic prescribing for those with acute respiratory infections (not confirmed bacterial disease) presenting to primary care (RR 0.77, 95%CI 0.69-0.86, 12 trials [10218 participants], moderate-certainty evidence). Although the performance characteristics of this test are insufficiently good to recommend its use in isolation, this evidence would suggest that this assay could play a useful role when integrated into a care pathway. Other biomarkers have not been proven to improve prescribing; one Swiss study using procalcitonin to guide antibiotic treatment for paediatric CAP did not find any benefit. However, this may well have been due to the fact that standard prescribing practices at these Swiss centres were already extremely good, as only 56% of children in the control group were given antibiotics. North American clinicians are much more liberal with antibiotic prescribing for CAP; unpublished MCH and CHEO data indicate that 99% of children diagnosed with CAP in the paediatric ED receive antibiotics, and American data show that most children diagnosed with CAP at outpatient clinics and EDs are also treated.

There have been very few trials investigating care pathways to improve antibiotic treatment of children with non-severe CAP in the ED. One cluster-randomized trial enrolled children with respiratory infections to assess the utility of an online digital calculator (developed to predict the likelihood of bacterial infections using many clinical and laboratory variables), where those randomized to the intervention arm were only prescribed antibiotics if the probability of bacterial disease was >10%; unfortunately, only 315/995 participants had CAP and there was no effect observed of the intervention on antibiotic use. Another study done in Italy using a different paediatric CAP care pathway did not even attempt to decrease unnecessary prescribing.

Overall, the effectiveness of care pathways will vary widely depending on how they are constructed and by what constitutes local standard of care. In the PIONEER pilot study that just finished enrolling at MCH, 100% of participants with CAP who received standard care received antibiotics, whereas only 53% of participants with CAP whose care was guided by the novel care pathway (the intervention of interest) were prescribed antibiotics within 14 days. The absolute benefit of our intervention may prove to be substantially larger than that reported for other stewardship interventions aiming to improve antimicrobial use for respiratory infections.

ELIGIBILITY:
Inclusion Criteria:

Children aged 6 month to 18 years presenting to the Emergency Department who are diagnosed with CAP and are well enough to be discharged home (i.e. 'non-severe' CAP) will be eligible. They must have a fever (on exam or by history) and at least one of:

* Tachypnoea measured at triage (>60 bpm for age <1, >50 for 1-2 years of age, >40bpm for 2-4 years of age, and >30bpm for >4 years of age)
* Cough on exam or by history
* Increased work of breathing on exam
* Auscultatory finding (focal crackles, bronchial breathing, etc.) consistent with CAP

Exclusion Criteria:

Children will be excluded if they have any of the following

* Cystic Fibrosis
* Anatomic Lung Disease
* Bronchiectasis
* Chronic Lung Disease requiring home oxygen or home ventilation
* Congenital heart Disease (requiring specific medical treatment or with exercise restrictions),
* History of repeated aspiration/velopharyngeal incompetence
* Malignancy
* Immunodeficiency (primary, acquired or iatrogenic)
* Pneumonia previously (clinically) diagnosed within the past month (that was presumed to have resolved prior to the episode prompting the current visit to the ED)
* Lung abscess within the past 6 months
* Children who present with ongoing fever after 4 days of amoxicillin, cefprozil, cefuroxime, levofloxacin, moxifloxacin or doxycycline are not eligible; as this duration of therapy with these drugs would normally be sufficient to treat bacterial CAP, a different approach would be required (ie. the care pathway as written might not be appropriate).
* Children will not be eligible to participate more than once

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 698 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2029-12-31 (Estimated); Study Completion 2030-06-30 (Estimated)

PRIMARY OUTCOMES:
Antibiotic use for CAP or respiratory tract infection before day 7 post-enrolment | From enrollment to 7 days post enrollment
  The proportion of patients who receive antibiotics.
Early clinical response (ECR, clinical improvement in symptoms and lack of requirement for additional antibacterials as measured at day 4). | From enrollment to day 4
  At baseline/enrollment, caregivers will be asked to rank all of the child's symptoms (work of breathing, dyspnoea [for children over the age of 7], oral intake, and activity level) as compared to normal. These will be categorized as the following: "same as normal", "a little worse than normal", and "a lot worse than normal". At the day 4, and day 15 follow-ups, caregivers will be asked to rank the child's symptoms as compared to the previous visit. These will be categorized as the following: "worse", "about the same", "a little better", "a lot better". Clinical response requires at least "a little better" for any symptom that was not "same as normal" at baseline. Dyspnoea will be self-reported in children over the age of seven. For those under seven, dyspnoea will not be reported.

SECONDARY OUTCOMES:
Ordinal outcome variable | From enrollment to end of 30 day follow up
  This variable will include early clinical response, drug adverse events, and hospitalization to generate an ordinal outcome variable with ranks 1-8. Ranks 1-3 have ECR being met with no AEs; mild-moderate AEs; and severe AEs, respectively. Ranks 4-6 are associated with NOT achieving ECR with no AEs; mild-moderate AEs; and severe AEs, respectively. Rank 7 is no ECR plus hospitalization with no AEs, and rank 8 is no ECR with hospitalization and any AE.
Time to resolution of both fever and iincreases work of breathing | From enrollment to end of 30 day follow up
Late clinical response | From enrollment to day 15
  Defined same as early clinical response but measured at day 15 as compared to day 4
Proportion of participants with antibiotic use specifically for CAP or respiratory tract infection before day 30 | From enrollment to end of 30 day follow up
Hospitalization for CAP before day 30 | From enrollment to end of 30 day follow up
The occurrence of drug-related adverse events | From enrollment to end of 30 day follow up
The occurrence of severe drug-related adverse events | From enrollment to end of 30 day follow up
Unscheduled ED or urgent care visits before day 15 | From enrollment to day 15
The development of complicated CAP (i.e. pleural effusion/empyaema) before day 15 | From enrollment to day 15
The number of days that participants miss school/daycare before day 15 | From enrollment to day 15
The acceptability of the care plan from the caregiver's perspective on day 0 and day 30 | From enrollment to end of 30 day follow up
  Questionnaire given to parents to assess the acceptability of the care plan will be completed on day 30. This is a 6-point Likert scale ranging from 'extremely satisfied' to 'not at all satisfied'
The number of days that participant's caregivers have work disrupted before day 15 | From enrollment to day 15

CONTACTS AND LOCATIONS:
Locations (6):
- Canada (6):
  - Alberta Children's hospital, Calgary, Alberta
  - Stollery Children's Hospital, Edmonton, Alberta
  - BC Children's Hospital, Vancouver, British Columbia
  - McMaster Children's Hospital, Hamilton, Ontario
  - Children's Hospital of Eastern Ontario (CHEO), Ottawa, Ontario
  - The Hospital for Sick Children, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No